CLINICAL TRIAL: NCT00378001
Title: A Prospective, Multicenter, Investigator Blinded, Randomized, Concurrent Control Study of Efficacy and Tolerability of Two FSH Preparations (Fostimon® Versus Gonal-F®) in Women Undergoing IVF
Brief Title: Clinical Efficacy and Tolerability of Two FSH Preparations (Human FSH Versus rFSH - Follitropin Alpha) in Women Undergoing IVF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03CHUS/FSH03
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Infertility
Keywords: Infertility, FSH, IVF, Ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — follitropin alfa

INTERVENTIONS:
Drug: FSH-IBSA
Drug: GONAL-F

SUMMARY:
The purpose of the study is to evaluate the clinical efficacy and general tolerability of two different subcutaneous FSH preparations (Fostimon®, IBSA vs Gonal-F®, Serono Inc.) when administered to patients undergoing controlled ovarian stimulation for IVF.

DETAILED DESCRIPTION:
This is a prospective, multicenter, investigator blinded, randomized, concurrent control, phase III clinical trial. Patients meeting the eligibility requirements of the study will be randomly assigned to receive either the test drug (Fostimon®, IBSA) or the reference drug (Gonal-F®, Serono Inc.). Investigators will be blinded by not allowing them to have any contact with the study medications (supplied in boxes labeled in a manner that does not reveal the content of the boxes), and requesting that patients do not make any statements to the investigator that might indicate the treatment to which they were assigned. Equivalence testing with regard to the primary outcome variable will establish whether the two treatments are indeed similarly effective.

ELIGIBILITY:
Inclusion Criteria:

* >/=18 and <40 years old;

  * BMI between 18 and 30 kg/m2;
  * less than 3 previously completed IVF cycles (i.e. completed cycle = egg recovery);
  * basal FSH <10 IU/L and E2 <80 pg/mL;
  * Within 12 months of the beginning of the study, uterine cavity consistent with expected normal function as assessed through a hysterosalpingogram, sonohysterogram, or hysteroscopic examination;
  * >10 antral follicles 2-10 mm in size;
  * Normal or clinically insignificant hematology and blood chemistry values. TSH levels must be within the normal limits for the testing laboratory, or the patient should be euthyroid as determined by the investigator (e.g. normal free thyroxine). TSH can be low secondary to exogenous thyroid medication where patient is euthyroid;
  * Able and willing to sign the Patient Consent Form and adhere to the study visitation schedule.

Exclusion Criteria:

* · age <18 and >/=40 years;

  * primary ovarian failure or women known as poor responders (i.e. requiring more than 300 IU of FSH as a starting dose in previous treatment cycles or having less than 3 oocytes retrieved, or with an E2 serum concentration <1800 pmol/L/500pg/mL);
  * prior ovarian hyperstimulation syndrome (OHSS), polycystic ovarian syndrome that would normally be started at a lower FSH dose than is initially required by the study (i.e. 300 IU), or likely intolerance to even two days of 300 IU FSH.
  * one or both ovaries inaccessible for oocyte retrieval;
  * ovarian cysts >20 mm;
  * hydrosalpinx that have not been surgically removed or ligated;
  * stage 3 or 4 endometriosis;
  * oocyte donation;
  * implantation of previously frozen embryos;
  * patients affected by pathologies associated with any contraindication of being pregnant;
  * hypersensitivity to the study medication;
  * abnormal bleeding of undetermined origin;
  * uncontrolled thyroid or adrenal dysfunction;
  * neoplasias;
  * severe impairment of renal and/or hepatic function;
  * use of concomitant medications that might interfere with study evaluations (e.g. nonstudy hormonal medications, prostaglandin inhibitors, psychotropic agents).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the total number of oocytes retrieved.

SECONDARY OUTCOMES:
Total FSH dose (IUs);number of days of FSH stimulation and stimulation duration;number of follicles >14 mm on the day of hCG injection;
17-β estradiol (E2) serum concentration on the day of hCG injection;cancellation rate with reasons;
Fertilization rate: number of 2PN (or already cleaved) embryos;
Total number of embryos,number transferred, frozen and discarded;implantation rate;number of transferred embryos; clinical pregnancy rate, per stimulated cycle, per oocyte retrieval and per embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Baker, MD, Principal Investigator — Fertility Physicians of Northern California; Victor Y Fujimoto, MD, Principal Investigator — UCSF In Vitro Fertilization; L. Michael Kettel, MD, Principal Investigator — San Diego Fertility Center; Michael R Soules, MD, Principal Investigator — Seattle Reproductive Medicine
Locations (4):
- United States (4):
  - Fertility Physicians of Northern California, Palo Alto, California
  - San Diego Fertility Center, San Diego, California
  - UCSF In Vitro Fertilization, San Francisco, California
  - Seattle Reproductive Medicine, Seattle, Washington

REFERENCES:
- [Background] Templeton A, Morris JK. Reducing the risk of multiple births by transfer of two embryos after in vitro fertilization. N Engl J Med. 1998 Aug 27;339(9):573-7. doi: 10.1056/NEJM199808273390901. PMID 9718375
- [Background] Porter RN, Smith W, Craft IL, Abdulwahid NA, Jacobs HS. Induction of ovulation for in-vitro fertilisation using buserelin and gonadotropins. Lancet. 1984 Dec 1;2(8414):1284-5. doi: 10.1016/s0140-6736(84)92840-x. No abstract available. PMID 6150318
- [Background] Loumaye E. The control of endogenous secretion of LH by gonadotrophin-releasing hormone agonists during ovarian hyperstimulation for in-vitro fertilization and embryo transfer. Hum Reprod. 1990 May;5(4):357-76. doi: 10.1093/oxfordjournals.humrep.a137105. No abstract available. PMID 2193939
- [Background] Hughes EG, Fedorkow DM, Daya S, Sagle MA, Van de Koppel P, Collins JA. The routine use of gonadotropin-releasing hormone agonists prior to in vitro fertilization and gamete intrafallopian transfer: a meta-analysis of randomized controlled trials. Fertil Steril. 1992 Nov;58(5):888-96. doi: 10.1016/s0015-0282(16)55430-2. PMID 1426372
- [Background] Smitz J, Devroey P, Braeckmans P, Camus M, Khan I, Staessen C, Van Waesberghe L, Wisanto A, Van Steirteghem AC. Management of failed cycles in an IVF/GIFT programme with the combination of a GnRH analogue and HMG. Hum Reprod. 1987 May;2(4):309-14. doi: 10.1093/oxfordjournals.humrep.a136540. PMID 3114314
- [Background] Giudice E, Crisci C, Eshkol A, Papoian R. Composition of commercial gonadotrophin preparations extracted from human post-menopausal urine: characterization of non-gonadotrophin proteins. Hum Reprod. 1994 Dec;9(12):2291-9. doi: 10.1093/oxfordjournals.humrep.a138440. PMID 7714147
- [Background] Howles CM, Loumaye E, Giroud D, Luyet G. Multiple follicular development and ovarian steroidogenesis following subcutaneous administration of a highly purified urinary FSH preparation in pituitary desensitized women undergoing IVF: a multicentre European phase III study. Hum Reprod. 1994 Mar;9(3):424-30. doi: 10.1093/oxfordjournals.humrep.a138522. PMID 8006130
- [Background] Wikland M, Borg J, Hamberger L, Svalander P. Simplification of IVF: minimal monitoring and the use of subcutaneous highly purified FSH administration for ovulation induction. Hum Reprod. 1994 Aug;9(8):1430-6. doi: 10.1093/oxfordjournals.humrep.a138724. PMID 7989500
- [Background] Daya S, Gunby J, Hughes EG, Collins JA, Sagle MA. Follicle-stimulating hormone versus human menopausal gonadotropin for in vitro fertilization cycles: a meta-analysis. Fertil Steril. 1995 Aug;64(2):347-54. PMID 7615113
- [Background] Golan A, Ron-el R, Herman A, Soffer Y, Weinraub Z, Caspi E. Ovarian hyperstimulation syndrome: an update review. Obstet Gynecol Surv. 1989 Jun;44(6):430-40. doi: 10.1097/00006254-198906000-00004. No abstract available. PMID 2660037